CLINICAL TRIAL: NCT06624618
Title: Rapid Molecular Detection of Sepsis in Whole Blood
Brief Title: Rapid Molecular Diagnosis of Sepsis in the Intensive Care Unit
Acronym: RADOS
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Health Holland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0344
Record Dates: First submitted 2024-04-30; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Sepsis; Bloodstream Infection
Keywords: Culture-free; Whole blood; Molecular diagnosis; Sepsis; Bloodstream infection; Bacterial DNA
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Lysed whole blood samples from which microbial DNA has been isolated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Rapid diagnosis of sepsis is crucial for treatment and survival. Currently, blood culture takes 48 hours-5 days to complete. After starting antimicrobial treatment blood culture results are not reliable. As a result, empirical broad spectrum antimicrobial therapy is mostly used. This implies possible antimicrobial over- or under treatment which is associated with increased antimicrobial resistance development. Early identification of the causative pathogen of sepsis will therefore have a major impact on the adequate treatment and reduction of high mortality rates. To date, there is not a single molecular diagnostic test available on the market to detect all putative causative bacterial pathogens of sepsis. In this study, the investigators will develop and validate a completely new molecular sepsis approach based on pathogen DNA detection, as an alternative to culture.

ELIGIBILITY:
Inclusion Criteria:

-Patients are included when routine blood cultures are ordered for diagnosis of bloodstream infections.

Exclusion Criteria:

-N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the Intensive Care Unit (ICU) of Maastricht University Medical Center (MUMC) are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Development and validation of rapid diagnostics tests for detection of bacterial DNA in sepsis | 2 years
  The tests will report presence of bacterial DNA by giving a specific bacterial species name.
Patterns of bacterial DNA dynamics over time | 2 years
  Use of species-specific qPCR primers (either from existing sepsis literature or to be designed) to quantify the DNA load at at least 3 different time points during an infectious episode. Comparison of these loads with infectious parameters used for routine diagnostics and with antibiotic use.

SECONDARY OUTCOMES:
Distinguishing between the causative pathogen and contamination by a physician evaluation panel, both for the current gold standard (blood cultures) and the results of new microbiological tests for detecting sepsis pathogens | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands